CLINICAL TRIAL: NCT02310022
Title: A Pharmacokinetic and Pharmacodynamic Study of Two Formulations of Omega-3 One Gram Capsules After Single and Multi-Dose Administrations Under Fed Conditions
Brief Title: A PK and PD Study of Two Formulations of Omega-3 One Gram Capsules
Acronym: PK/PD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Matinas Biopharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MB-70001
Record Dates: First submitted 2014-11-14; First posted 2014-12-05 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — MAT9001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Omega 3 (Experimental): 4g (4 capsules) once a day, administered with food Other name MAT9001
  Interventions: Drug: Drug Omega 3
- Drug Omega 3 Comparator (Active Comparator): 4g (4 capsules) once a day, administered with food Other name Omega 3 Active Comparator
  Interventions: Drug: Drug Omega-3 Comparator

INTERVENTIONS:
Drug: Drug Omega 3 — 4 g (4 capsules) once a day, administered with food
  Other Names: MAT9001
  Arms: Drug Omega 3
Drug: Drug Omega-3 Comparator — 4 g (4 capsules) once a day, administered with food
  Other Names: Active Comparator
  Arms: Drug Omega 3 Comparator

SUMMARY:
Comparative bioavailability and pharmacodynamics effects of MAT9001 versus an active omega-3 medication comparator.

DETAILED DESCRIPTION:
The primary objective is to determine the comparative bioavailability and pharmacodynamics effects of single and multiple doses of MAT9001 versus an active omega-3 medication comparator.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfil all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

1. Adult male or female subject, 18-70 years of age, inclusive.
2. Light- or non-smoking, male and female subjects, 18 to 70 years of age. Note: subjects that regularly smoke greater than 10 cigarettes per day will not be considered light-smokers and should not be included. Additionally, the use of any cigars, pipes, vapor inhalers or any other tobacco containing product is prohibited within 6 months prior to drug administration.
3. Body mass index (BMI) ≥ 19 and ≤ 40 (kg/m2).
4. No clinically significant findings in vital signs measurements. The acceptable range for seated systolic blood pressure is 90-150 mmHg and for diastolic blood pressure is 50-95 mmHg.
5. No clinically significant abnormal laboratory values that, in the opinion of the investigator, would compromise the subject's safety or the integrity of the study results.
6. Either have: elevated triglyceride levels (2.26 to 4.52 mmol/L [200 to 400 mg/dL]), or · triglyceride levels 2.26 to 3.95 mmol/L (200 to 350 mg/dL) and are on stable statin therapy.
7. Total cholesterol levels ≤ 7.75 mmol/L (≤ 300 mg/dL).
8. Hemoglobin ≥ 135 g/L for males or ≥ 120 g/L for females at screening.
9. No clinically significant findings in a 12-lead electrocardiogram (ECG)
10. Have no significant diseases.
11. Willing to use an acceptable, effective method of contraception.
12. Be informed of the nature of the study and give written consent prior to any study procedure.
13. Have no clinically significant findings from a physical examination.

Exclusion Criteria:

Subjects may be excluded from the study if there is evidence of any of the following criteria at screening, check-in, or at any time during the study, as appropriate:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurological, or psychiatric disease in the opinion of the PI.
2. Personal or familial history of bleeding disorder(s), thromboembolic disease, clinical GI bleeding, or any history of GI surgery except uncomplicated appendectomy or cholecystectomy, or colorectal surgery for polyps, nonmalignant tumors, or diverticula.
3. Positive urine drug/alcohol testing at screening or check-in.
4. Positive result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
5. History or presence of alcoholism or drug abuse within the past 2 years.
6. Known sensitivity or allergy to fish, shellfish, gelatin or omega-3 products.
7. Subject is a female who is pregnant or lactating.
8. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to drug administration
9. Donation of blood or significant blood loss within 56 days prior to check- in.
10. Participation in another clinical trial within 30 days prior drug administration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Bioavailability comparison after single and multiple doses over a 24 hour period at day 1 and day 14 | 14 Days
  Area under the plasma concentration curve versus time curve (AUC0-tau) versus time curve (AUC0-tau) for both treatments measured over the 24 hour period on day 1 and day 14 [ Time Frame: 14 days ]

SECONDARY OUTCOMES:
Comparison of baseline changes of triglycerides and other related lipid protein parameter levels over 14 days | 14 Days
  To compare the change from baseline triglyceride and other related lipid/lipoprotein parameter levels between:· MAT9001 and an active omega-3 medication comparator; after multi-dose administrations in subjects under fed conditions

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, MD, Study Director — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Reserach Inc, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Maki KC, Bobotas G, Dicklin MR, Huebner M, Keane WF. Effects of MAT9001 containing eicosapentaenoic acid and docosapentaenoic acid, compared to eicosapentaenoic acid ethyl esters, on triglycerides, lipoprotein cholesterol, and related variables. J Clin Lipidol. 2017 Jan-Feb;11(1):102-109. doi: 10.1016/j.jacl.2016.10.010. Epub 2016 Oct 18. PMID 28391875